CLINICAL TRIAL: NCT04049773
Title: Fatigue in Chronic Haemodialysis Patients: an Experience Sampling Method Study
Acronym: FatHoM
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: METCZ20190078
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-07

CONDITIONS: Fatigue; End Stage Renal Disease
Keywords: fatigue; haemodialysis; ecological momentary assessment
MeSH Terms: conditions — Fatigue; Kidney Failure, Chronic | interventions — Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Procedure: haemodialysis — haemodialysis, thrice weekly in-center

SUMMARY:
To investigate the course and diurnal change of fatigue symptoms and haemodialysis related symptoms in chronic haemodialysis patients, its relation to haemodialysis treatment and the association with other factors by implementing an ecological momentary assessment procedure incorporated in a webapplication.

DETAILED DESCRIPTION:
The course and diurnal change of fatigue symptoms in the daily life of chronic haemodialysis (HD) patients, its relation to haemodialysis treatment and the association with other factors such as mood, activities, location and social context will be evaluated during 7 consecutive days by using an ecological momentary assessment (EMA) procedure, incorporated into a webapplication. Using an EMA procedure will more accurately represent fatigue symptoms and its relation to other factors in the daily life of chronic HD patients compared to conventional measurement instruments (i.e. questionnaires evaluating fatigue over a period of a week or more, which are therefore liable to a recall bias).

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease requiring chronic haemodialysis treatment currently being treated for at least 6 months.
* Good understanding of Dutch based on clinical judgment (since the web-application is only available in the Dutch language).

Exclusion Criteria:

* The participant cannot independently handle the web-application based on clinical judgment.
* Dementia or insufficient cognitive skills to handle the web-application based on clinical judgement by the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: secondary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in fatigue symptoms throughout the day | 7 consecutive days
  self-reported fatigue intensity on a 7-point Likert scale (from 1 "not fatigued" to 7 "very fatigued") at ten occasions randomly throughout the day.

SECONDARY OUTCOMES:
Change in fatigue symptoms (primary outcome) and its association with mood | 7 consecutive days
  Questions with respect to mood are evaluated on a 7-point Likert scale (from 1 '"not at all" to 7"very much").
Change in fatigue symptoms (primary outcome) and its association with location, activities and social context | 7 consecutive days
  Location, social context and activities related questions are provided in a multiple-choice format.
Change in haemodialysis related symptoms (such as muscle cramps, itch, bone pain, headache) throughout the day | 7 consecutive days
  Self-reported intensity of the above-mentioned symptoms on a 7-point Likert scale (from 1 "not at all" to 7 "very much") at ten occasions randomly throughout the day.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Stifft, MD, Principal Investigator — Zuyderland MC; Caroline M van Heugten, PhD, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - ZuyderlandMC, Heerlen, Limburg
  - ZuyderlandMC, Sittard, Limburg

IPD SHARING:
Plan to Share IPD: No